CLINICAL TRIAL: NCT01467700
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Once a Day, TAK-375 (Ramelteon) Tablet for Sublingual Administration (TAK-375SL Tablet) in the Treatment of Acute Depressive Episodes Associated With Bipolar I Disorder in Adult Patients Who Are on Lithium and/or Valproate
Brief Title: Efficacy and Safety of Ramelteon Sublingual in Adult Patients With Acute Depressive Episodes Associated With Bipolar I Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; No Safety Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375SL_201; U1111-1122-7380 (Registry Identifier: WHO)
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Acute Depressive Episode
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ramelteon SL 0.1 mg (Experimental): Ramelteon SL 0.1 mg, tablets, sublingual (SL) [dissolved under the tongue], once daily (QD), every night at bedtime for up to 8 weeks.
  Interventions: Drug: Ramelteon SL
- Ramelteon SL 0.4 mg (Experimental): Ramelteon SL 0.4 mg, tablets, sublingual, once daily, every night at bedtime for up to 8 weeks.
  Interventions: Drug: Ramelteon SL
- Ramelteon SL 0.8 mg (Experimental): Ramelteon SL 0.8 mg tablets, sublingual, once daily, every night at bedtime for up to 8 weeks.
  Interventions: Drug: Ramelteon SL
- Placebo (Placebo Comparator): Ramelteon SL placebo-matching, tablets, sublingual, once daily, every night at bedtime for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon SL — Ramelteon SL tablets
  Other Names: TAK-375SL
  Arms: Ramelteon SL 0.1 mg; Ramelteon SL 0.4 mg; Ramelteon SL 0.8 mg
Drug: Placebo — Ramelteon placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Ramelteon, once daily (QD), sublingual (SL), in adult participants with acute depressive episodes associated with Bipolar I disorder.

DETAILED DESCRIPTION:
Ramelteon sublingual formulation is being developed by Takeda Pharmaceutical Company Limited for maintenance therapy of Bipolar I disorder.

Participants will be seen twice during the first week of treatment, weekly during the first 2 weeks of treatment and then every 2 weeks up to the end of the 8-week treatment period. Participants who complete the 8-week treatment period will have a follow-up visit approximately seven days after the last visit. A safety follow-up phone call will be made 30 days after completion of the 8-week treatment period.

Based on the recommendation of the Independent Data Monitoring Committee which determined that the study data had met pre-determined criteria for futility, Takeda has made a decision to terminate the study. No safety concerns were identified by the Independent Data Monitoring Committee

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a man or woman aged between 18 and 75 years, inclusive.
4. The participant suffers from Bipolar I Disorder, Most Recent Episode Depressed as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.5x) and confirmed by the Structured Clinical Interview for DSM Disorders (SCID).
5. The reported duration of the current Major Depressive Episode (MDE) is at least four weeks and less than 6 months.
6. The participant has a Young Mania Rating Scale (YMRS) score of ≤10 both at the Screening and Baseline visits.
7. The participant has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥24 at the Screening and Baseline Visits.
8. The participant has a Clinical Global Impression Scale - Severity (CGI-S) score of ≥4 at the Screening and Baseline Visits.
9. Hamilton Rating Scale for Anxiety (HAM-A) score is ≤21 at Screening and Baseline visits.
10. The participant has a lithium and/or valproate levels within therapeutic range (0.6 - 1.2 mEq/L for lithium or 50-125 mcg/ml for valproate) at screening. If the patient does not have a lithium and/or valproate level within therapeutic range at screening, they must have a lithium and/or valproate levels within the therapeutic range between Day - 15 to Day -30 of screening.
11. A female participant of childbearing potential who is sexually active and agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose.
12. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent through the duration of the study and for 30 days after the last dose.

Exclusion Criteria:

1. The participant has received any investigational compound <30 days before Screening or 5 half-lives prior to Screening.
2. The participant has received ramelteon in a previous clinical study or has ever used ramelteon.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
4. The participant has one or more of the following:

   * Any current psychiatric disorder other than Bipolar I Disorder, Most Recent Episode Depressed as defined in the DSM-IV-TR, as assessed by the SCID.
   * Current or history of: schizophrenia, unipolar depression with psychotic features, bipolar depression with psychotic features, any other psychotic disorder (with the exception of psychosis associated with a manic episode), mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   * Current diagnosis or history of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at least one year from the day of screening. (Participant must also have negative urine drug screen prior to Baseline).
   * Presence or history of a clinically significant neurological disorder (including epilepsy).
   * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
   * Any Axis II disorder that might compromise the study.
   * History of Rapid Cycling Bipolar Disorder: Patients who have more than 8 episodes of mood disorder per year.
5. The participant experienced the first episode of mood disorder after the age of 65 years.
6. The current depressive symptoms of the participant are considered by the investigator to have been resistant to 2 adequate treatment trials with any of the mood stabilizers (specifically started to treat the current depressive episode) and/or antidepressant medications of at least 6 weeks duration each.
7. The participant is on any other psychotropic medications except for lithium (serum levels 0.8 to mEq/L) or valproate (serum levels 50 to 125 mcg/ml) at the Screening visit.
8. The participant is on lithium and/or valproate for less than 30 days prior to screening.
9. If the participant is on antidepressant medications and/or antipsychotic medications (used as a mood stabilizer) and the patient is considered appropriate by the PI, these medications must be washed out for at least 2 weeks prior to the Screening visit.
10. The participant has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
11. The participant has started receiving formal cognitive or behavioral therapy, systematic psychotherapy within 30 days prior to screening or plans to initiate such therapy during the study.
12. The participant has a significant risk of suicide according to the investigator's clinical judgment or has a score ≥ 5 on item 10 (suicidal thoughts) of the MADRS or has made a suicide attempt in the previous 6 months.
13. The participant has taken or is anticipated that the participant will take at least 1 of the disallowed concomitant medications.
14. The participant has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, hematological, infectious, dermatological disorder or metabolic disturbance as determined by Investigator.
15. The participant has a history or current diagnosis of Fibromyalgia, Chronic Fatigue Syndrome, Chronic Pain Syndrome or Sleep apnea.
16. The participant has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin.
17. The participant has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant; or the participant has any of the following values at the Screening Visit:

    * A serum creatinine value >1.5 times the upper limits of normal (xULN).
    * A serum total bilirubin value >1.5 xULN.
    * A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 xULN.
18. The participant has glycosylated hemoglobin (HbA1C) ≥7% at baseline and no prior diagnosis of diabetes and/or treatment for diabetes. NOTE: Participants with known diabetes are not excluded.
19. The participant has a thyroid stimulating hormone (TSH) value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator. If TSH is outside the normal range, a free T4 will be obtained.
20. The participant has clinically significant abnormal vital signs as determined by the investigator.
21. The participant has an abnormal electrocardiogram (ECG) as determined by the central reader and confirmed as clinically significant by the investigator.
22. The participant has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
23. The participant, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (160):
- United States (140):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Fayetteville, Arkansas
  - Little Rock, Arkansas
  - Bellflower, California
  - Costa Mesa, California
  - Garden Grove, California
  - Harbor City, California
  - Huntington Park, California
  - Irvine, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Murrieta, California
  - National City, California
  - Oceanside, California
  - Orange, California
  - Paramount, California
  - Rancho Cucamonga, California
  - Redondo Beach, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - San Jose, California
  - San Ramon, California
  - Sherman Oaks, California
  - Torrance, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Coral Gables, Florida
  - Coral Springs, Florida
  - Edgewater, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Lakes, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - East Point, Georgia
  - Smyrna, Georgia
  - Suwanee, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Gurnee, Illinois
  - Hoffman Estates, Illinois
  - Libertyville, Illinois
  - Skokie, Illinois
  - Brownsburg, Indiana
  - Manhattan, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Bloomfield Hills, Michigan
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Flowood, Mississippi
  - Hazelwood, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Cherry Hill, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Cedarhurst, New York
  - Fresh Meadows, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Columbiana, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - McMurray, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Lincoln, Rhode Island
  - Columbia, South Carolina
  - Greer, South Carolina
  - Old Point Station, South Carolina
  - Clarksville, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Bellaire, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Nassau Bay, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Kirkland, Washington
  - Richland, Washington
  - Seattle, Washington
  - Clarksburg, West Virginia
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Mendoza
  - Santa Fe
- Chile (4):
  - Antofagasta
  - Arauco
  - Elqui
  - Santiago
- Colombia (4):
  - Bello, Antioquia
  - Antioquia
  - Barranquilla
  - Bogotá
- Mexico (8):
  - Mexicali, Estado de Baja California
  - León, Guanajuato
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - San Lucas, Tepetlacalco
  - Mérida, Yucatán
  - México
  - San Luis Potosí City

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 98 investigative sites in Argentina, Chile, Colombia, Mexico and the United States 12 December 2011 (first participant signed the informed consent form) to 10 March 2015.
Pre-assignment Details: Participants with a diagnosis of acute depressive episode were enrolled equally in 1 of 4 treatment groups, once a day placebo, ramelteon [TAK-375 SL (sublingual)] 0.1 mg, 0.4 mg or 0.8 mg.
Groups:
- Placebo: Ramelteon SL placebo-matching, tablets, sublingual (SL) [dissolved under the tongue], once daily, every night at bedtime for up to 8 weeks.
- Ramelteon SL 0.1 mg: Ramelteon SL 0.1 mg, tablets, SL, once daily (QD), every night at bedtime for up to 8 weeks.
- Ramelteon SL 0.4 mg: Ramelteon SL 0.4 mg, tablets, SL, once daily, every night at bedtime for up to 8 weeks.
- Ramelteon SL 0.8 mg: Ramelteon SL 0.8 mg tablets, SL, once daily, every night at bedtime for up to 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Started | 115 | 128 | 124 | 123
Safety Set - Received Treatment | 115 | 127 | 124 | 123
Completed | 86 | 100 | 97 | 96
Not Completed | 29 | 28 | 27 | 27
Not completed — Pretreatment Event or Adverse Event | 6 | 4 | 2 | 3
Not completed — Major Protocol Deviation | 3 | 3 | 2 | 3
Not completed — Lost to Follow-up | 6 | 5 | 2 | 3
Not completed — Voluntary Withdrawal | 5 | 7 | 6 | 2
Not completed — Study Termination | 6 | 5 | 10 | 7
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 1
Not completed — Reason not Specified | 1 | 3 | 2 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg | Total
Number analyzed (Participants) | 115 | 128 | 124 | 123 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.95 (10.867) | 43.01 (11.998) | 42.96 (13.211) | 43.97 (10.243) | 43.69 (11.646)
Age, Customized [Number; unit: participants]
  <=50 Years | 85 | 92 | 88 | 97 | 362
  >50 Years | 30 | 36 | 36 | 26 | 128
Age, Customized [Number; unit: participants]
  <=65 years | 111 | 126 | 119 | 121 | 477
  >65 Years | 4 | 2 | 5 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 71 | 78 | 69 | 292
  Male | 41 | 57 | 46 | 54 | 198
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 36 | 38 | 35 | 37 | 146
  Non-Hispanic and Non-Latino | 79 | 90 | 89 | 86 | 344
Race/Ethnicity, Customized [Number; unit: participants]
  White | 76 | 81 | 85 | 79 | 321
  Black | 29 | 42 | 32 | 38 | 141
  Asian | 3 | 0 | 2 | 0 | 5
  American Indian or Alaska Native | 5 | 3 | 0 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 3
  Multiple | 1 | 2 | 4 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 85 | 97 | 95 | 94 | 371
  Argentina | 12 | 11 | 11 | 11 | 45
  Chile | 5 | 5 | 6 | 3 | 19
  Colombia | 3 | 3 | 1 | 3 | 10
  Mexico | 10 | 12 | 11 | 12 | 45
Height [Mean (Standard Deviation); unit: cm] | 166.93 (10.345) | 169.00 (9.937) | 167.22 (9.677) | 168.15 (10.590) | 167.85 (10.139)
Weight [Mean (Standard Deviation); unit: kg] | 85.44 (20.034) | 87.58 (21.555) | 85.09 (20.873) | 86.69 (21.535) | 86.22 (20.989)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated using the weight collected at the first screening visit: BMI=weight(kg)/[height(m)]^2.
  kg/m^2 | 30.62 (6.778) | 30.63 (7.254) | 30.37 (6.808) | 30.61 (6.825) | 30.56 (6.904)
Smoking Classification [Number; unit: participants]
  Participant Has Never Smoked | 47 | 55 | 49 | 45 | 196
  Participant is a Current Smoker | 50 | 58 | 58 | 58 | 224
  Participant is an Ex-smoker | 18 | 15 | 17 | 20 | 70
Participant Drinking Status [Number; unit: participants]
  Has Never Drunk | 52 | 41 | 45 | 49 | 187
  Ex-Drinker | 25 | 36 | 28 | 37 | 126
  Current Drinker | 22 | 34 | 33 | 25 | 114
  Missing | 16 | 17 | 18 | 12 | 63
If Drinker, Amount Consumed [Number; unit: participants] — Only participants with drinking status Current Drinker are accounted for: N=22, 34, 33, 25 in each treatment arm, respectively.
  participants
    < 4 drinks per day | 22 | 34 | 33 | 25 | 114
    >= 4 drinks per day | 0 | 0 | 0 | 0 | 0
Does Participant Consume Caffeine? [Number; unit: participants]
  Yes | 77 | 84 | 83 | 81 | 325
  No | 22 | 27 | 23 | 30 | 102
  Missing | 16 | 17 | 18 | 12 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: The change between MADRS score at week 6 relative to Baseline. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement. A mixed measures repeated measures (MMRM) model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: Participants from full analysis set (FAS), all randomized participants who, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary efficacy, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Ramelteon SL 0.4 mg: Ramelteon SL 0.4 mg, tablets, SL, once daily, every night at bedtime for up to 8 weeks,
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 103
score on a scale | -14.5 (0.94) | -14.4 (0.89) | -11.8 (0.91) | -14.8 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Ramelteon SL 0.1 mg; Test type: Superiority or Other; p = 0.518, Mixed Models Analysis — P-values were from an MMRM model with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis; LS Mean Difference = 0.1, 98% CI 2-sided [-2.9 to 3.1], Standard Error of Mean 1.28
Statistical Analysis 2: Comparison: Placebo vs Ramelteon SL 0.4 mg; Test type: Superiority or Other; p = 0.979, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 2.6, 98% CI 2-sided [-0.4 to 5.7], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Placebo vs Ramelteon SL 0.8 mg; Test type: Superiority or Other; p = 0.400, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.3, 99% CI 2-sided [-3.7 to 3.0], Standard Error of Mean 1.29

2. Secondary Outcome: Change From Baseline in Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) Short Form Total Score at Week 6
Description: Q-LES-Q -SF is a self-administered, 16-item questionnaire to assess the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning, such as social relationships, living/housing, physical health, medication, and global satisfaction. The questionnaire consists of 16 items rated by the participants on a 5-point scale. Of these, 14 items are summed to produce a total quality of life score with a maximum of 70 points. In addition, there are two global items that are scored individually. These items rate satisfaction with study medication and overall life satisfaction. The questionnaire is usually scored as a percent of total possible score, with higher scores indicating better health status. A positive change from Baseline indicates improvement. A MMRM model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: Participants from FAS, all randomized participants who, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary efficacy, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: percent of maximum score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 82 | 95 | 85 | 93
percent of maximum score on a scale | 8.4 (1.67) | 13.1 (1.56) | 9.2 (1.61) | 14.8 (1.57)
Statistical Analysis 1: Comparison: Placebo vs Ramelteon SL 0.1 mg; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 4.7, 98% CI 2-sided [-0.5 to 9.9], Standard Error of Mean 2.22
Statistical Analysis 2: Comparison: Placebo vs Ramelteon SL 0.4 mg; Test type: Superiority or Other; p = 0.361, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.8, 98% CI 2-sided [-4.5 to 6.1], Standard Error of Mean 2.25
Statistical Analysis 3: Comparison: Placebo vs Ramelteon SL 0.8 mg; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 6.4, 99% CI 2-sided [0.6 to 12.1], Standard Error of Mean 2.23

3. Secondary Outcome: Percentage of Participants With MADRS Response at Week 6, With Response Defined as a ≥ 50% Decrease in the MADRS Total Score From Baseline
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 103
percentage of participants | 45.2 | 50.5 | 47.5 | 52.4

4. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Week 6
Description: The YMRS total score at week 6 relative to baseline. YMRS is a four item scale to assess manic symptoms, rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe), with 7 items rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe) with higher scores reflecting greater levels of mania. The YMRS total score is calculated as the sum of the 11 individual item scores and ranges from 0-60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement. A MMRM model was used for analyses with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 103
score on a scale | -0.9 (0.35) | -0.8 (0.33) | -0.7 (0.34) | -0.4 (0.34)

5. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I) Score at Week 6
Description: The CGI-I assesses the clinician's impression of the participant's state of mental illness improvement and consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on a seven-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change relative to baseline; 5=minimally worse; 6= much worse; 7=very much worse). Higher scores indicate greater severity of illness. A MMRM model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: 6 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 102
score on a scale | 2.6 (0.10) | 2.6 (0.10) | 2.8 (0.10) | 2.6 (0.10)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity (CGI-S) at Week 6
Description: The CGI-S at week 6 relative to Baseline. The CGI-S assesses the clinician's impression of the participant's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill). Higher scores indicate greater severity of illness. A MMRM model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 103
score on a scale | -1.3 (0.11) | -1.3 (0.10) | -1.1 (0.10) | -1.3 (0.10)

7. Secondary Outcome: Percentage of Participants With MADRS Remission at Week 6, With Remission Defined as a MADRS Total Score ≤10
Description: as for outcome 3
Time Frame: Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 93 | 109 | 101 | 103
percentage of participants | 30.1 | 36.7 | 31.7 | 35.9

8. Secondary Outcome: Change From Baseline in the Quick Inventory of Depressive Symptomatology - Self-Rated16 (QIDS-SR16) Total Score at Week 6
Description: The 16 item QIDS-SR16 version is designed to assess the severity of depressive symptoms. The QIDS-SR16 assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 4th edition, DSM-IV, to diagnose a major depressive episode. QIDS-SR16 assessment has been used to screen for depression and also to measure symptom severity. This scale is also used to distinguish response from remission, as well as to quantify between group treatments effects in open label and randomized controlled trials. The patient is asked to rate the severity and frequency of specific symptoms present over the last 7 days. The QIDS-SR16 total scores range from 0 to 27. Higher scores indicate greater severity of impairment. A negative change from Baseline indicates improvement. A MMRM model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 66 | 82 | 78 | 78
score on a scale | -6.1 (0.59) | -6.2 (0.54) | -4.3 (0.54) | -6.2 (0.55)

9. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 6
Description: The SDS comprises patient-rated items designed to measure the extent to which the subject's life is impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his or her (1) work, (2) social life or leisure activities, and (3) home life or family responsibilities, are impaired by his or her symptoms on 10-point visual analogue scales from 0 (not at all) to 10 (extremely) with a total score range from 0 to 30. Higher scores indicate greater severity of impairment. There are verbal descriptors for the points on the scales as well as numerical scores that provide more precise levels of the verbal descriptors. In addition, the SDS addresses the number of days lost and the number of days under-productive due to the symptoms. A negative change from Baseline indicates improvement. A MMRM model was used for analysis with baseline*week, pooled center, week, treatment, baseline, and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 92 | 109 | 100 | 102
score on a scale | -5.1 (0.71) | -6.8 (0.66) | -4.1 (0.67) | -5.7 (0.68)

ADVERSE EVENTS:
Time Frame: Approximately 30 days after the last dose of study drug (up to 12 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Serious Adverse Events (participants affected / at risk) | 4/115 | 5/127 | 3/124 | 1/123
Other Adverse Events (participants affected / at risk) | 10/115 | 17/127 | 19/124 | 19/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | Ramelteon SL 0.1 mg (N=127) | Ramelteon SL 0.4 mg (N=124) | Ramelteon SL 0.8 mg (N=123)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 4 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | Ramelteon SL 0.1 mg (N=127) | Ramelteon SL 0.4 mg (N=124) | Ramelteon SL 0.8 mg (N=123)
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 8 | 5
Nasopharyngitis (Infections and infestations) | 2 | 7 | 2 | 6
Headache (Nervous system disorders) | 8 | 3 | 6 | 6
Somnolence (Nervous system disorders) | 0 | 7 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.